CLINICAL TRIAL: NCT01546454
Title: Identification of the Menstrual Cycle-Associated Factors That Modulate Circulating Lipid Levels in Premenopausal Women
Brief Title: Relationship Between the Menstrual Cycle and Heart Disease in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Director, Women's Health Research Unit, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB8023
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Coronary Heart Disease
Keywords: Premenopausal women; coronary heart disease; menstrual cycle; lipids
MeSH Terms: conditions — Coronary Disease | interventions — ethinyl estradiol, levonorgestrel drug combination; Leuprolide; luprolide acetate gel depot; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-steroidal effects (Experimental): Natural menstrual cycle versus Estrogen/Progesterone replacement cycle. Interventions include leuprolide acetate to induce hypogonadism and estradiol and progesterone to replace hormone levels.
  Interventions: Drug: leuprolide acetate; Drug: Estradiol; Drug: Progesterone
- Contraceptive effects (Experimental): Oral contraceptive cycle versus Eligard treatment. Interventions include ethinyl estradiol-levonorgestrel combination and leuprolide acetate.
  Interventions: Drug: Ethinyl Estradiol-Levonorgestrel combination; Drug: leuprolide acetate
- Steroid effects (Experimental): Estrogen/Progesterone replacement cycle versus Eligard treatment. Interventions include leuprolide acetate, estradiol, and progesterone.
  Interventions: Drug: leuprolide acetate; Drug: Estradiol; Drug: Progesterone

INTERVENTIONS:
Drug: Ethinyl Estradiol-Levonorgestrel combination — 0.03 mg ethinyl estradiol, 0.15 mg levonorgestrel oral daily for 21 days
  Other Names: Portia 21; Portia 28
  Arms: Contraceptive effects
Drug: leuprolide acetate — single 22.5 mg subcutaneous depot suspension
  Other Names: Eligard
Drug: Estradiol — 0.05 to 0.3 mg transdermal daily for 26 days
  Other Names: Vivelle-Dot
  Arms: Non-steroidal effects; Steroid effects
Drug: Progesterone — 50 to 100 mg vaginal suppositories twice daily for 13 days
  Other Names: First-Progesterone VGS
  Arms: Non-steroidal effects; Steroid effects

SUMMARY:
Women who have regular menstrual cycles have a lower risk of heart disease than men of the same age or women who no longer have menstrual cycles. The purpose of this study is to help determine why the menstrual cycle causes a lower risk of heart disease. The investigators believe that the hormones (estradiol and progesterone) produced during the menstrual cycle, as well as the normal processes occurring in the follicle and corpus luteum (transformed follicle), change levels of "good" and "bad" cholesterol in the blood-stream. These levels of good and bad cholesterol are an important risk factor for heart disease. Therefore, our goal is to determine what effects each of these factors (estradiol, progesterone, follicle, corpus luteum) have on the levels of good and bad cholesterol in the woman's bloodstream. As many women take birth control pills, which contain synthetic forms of estradiol and progesterone that block ovulation and development of a corpus luteum, the investigators also want to determine what effect one common type of birth control pill has on levels of good and bad cholesterol.

DETAILED DESCRIPTION:
Premenopausal women are at a lower age-adjusted risk of coronary heart disease (CHD) than men or postmenopausal women. This decreased risk of CHD is likely due, in part, to the more favorable lipid profile observed in premenopausal women. The menstrual cycle is associated with the ovarian processes of follicular growth and ovulation, and corpus luteum (CL) development, function, and regression. The steroids estrogen (E2) and progesterone (P4) are secreted from the follicle and CL, which travel via the bloodstream to elicit their effects on target tissues. The production of E2 has been implicated as the menstrual cycle-associated factor underlying the favorable lipid profile as it is known to increase atheroprotective high density lipoprotein and decrease atherogenic low density lipoprotein. However, other factors may play a role such as direct ovarian metabolism of circulating lipids. Furthermore, the role of P4 is unclear and there is some evidence that it may inhibit the beneficial effects of E2. Therefore, we aim to determine the contributions of ovarian metabolism of lipids, independent of the effects of ovarian-derived E2 and P4, to the circulating lipid profile in premenopausal women. Also, we will determine the relationship between E2 and P4, both natural and synthetic forms found in hormonal oral contraceptives, on circulating lipids. With the recent controversial findings of the Women's Health Initiative, further evaluation of the factors underlying menstrual cycle protection from CHD is warranted. This study may have implications for the management of CHD and the use of hormonal therapies in women.

ELIGIBILITY:
Inclusion Criteria:

* Normal menstrual cycles of 25-35 days in length for at least previous 3 cycles
* 21-40 years of age
* BMI > 18, < 30
* Serum P4 > 9 ng/ml on single sample collected between days 18-25 of self-reported menstrual cycle
* Flexible schedule allowing morning blood draws on less than 48 hour notice
* In good general health
* Commit to remain on stable diet during study period (no changes to normal dietary habits)
* Commit to using non-hormonal contraceptive methods during study period except those prescribed in the experimental protocol
* No objections to taking study drugs

Exclusion Criteria:

* Oral contraceptive use or other hormone supplement within the preceding 2 months
* Long-acting hormonal contraceptive use in the past 12 months (e.g., Depo-Provera®)
* Contraindications to study drugs
* Current or past pregnancy within the previous 6 months or currently trying to conceive
* Desiring to conceive in the next 8 months
* Breastfeeding in the past 2 months
* Diagnosed Diabetes or Metabolic Syndrome
* Current or previous use of cholesterol lowering drugs within the preceding 12 months
* Diagnosed Polycystic Ovary Syndrome
* History of, or self-reported, substance abuse
* Smoker
* Previous infertility treatment excluding male factor issues
* Use of an investigational drug within the past 2 months

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Jensen, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Sciences University, Department of Obstetrics and Gynecology, Women's Health Research Unit, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled participant was lost to follow-up prior to receiving any interventions.
Period: Natural Menstrual Cycle
Arm/Group | All Study Participants
Started | 4
Completed | 4
Not Completed | 0
Period: Oral Contraceptive Cycle
Arm/Group | All Study Participants
Started | 4
Completed | 4
Not Completed | 0
Period: Eligard Treatment
Arm/Group | All Study Participants
Started | 4
Completed | 4
Not Completed | 0
Period: Estrogen/Progesterone Replacement Cycle
Arm/Group | All Study Participants
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy premenopausal women from the Portland, OR metro area
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Total to HDL Cholesterol Ratio
Time Frame: Entire Study
Measure: Mean (95% Confidence Interval); unit: Total to HDL Cholesterol Ratio
Arm/Group | Non-steroidal Effects | Contraceptive Effects | Steroid Effects
Number analyzed (Participants) | 4 | 4 | 4
Total to HDL Cholesterol Ratio | 0.146 [0.033 to 0.26] | 0.148 [-0.13 to 0.43] | -0.89 [-2.09 to 0.315]

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No